CLINICAL TRIAL: NCT06902064
Title: Efficacy and Mechanism of Transcranial Temporal Interference Stimulation (tTIS) in the Treatment of Adolescent Depression
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY20242385
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Adolescent; Depression - Major Depressive Disorder
Keywords: adolescent; depression; Transcranial temporal interference stimulation
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tTIS Group (Experimental): This group received 10 sessions of tTIS treatment, once a day, each session lasting approximately 30 minutes.
  Interventions: Device: Transcranial temporal interference stimulation
- Sham group (Sham Comparator): This group will receive 10 sessions of sham tTIS treatment, once a day, each session lasting approximately 30 minutes.
  Interventions: Device: sham tTIS

INTERVENTIONS:
Device: Transcranial temporal interference stimulation — Transcranial temporal interference stimulation (tTIS) is a novel neurostimulation technique that utilizes two or more electric fields of specific frequencies to modulate the oscillations of neurons at the desired spatial location in the brain. The physics of tTIS offers the advantage of non-invasively regulating deep brain structures and minimally stimulating the overlying cortex outside the selected target.
  Other Names: tTIS
  Arms: tTIS Group
Device: sham tTIS — The sham tTIS is enabled by checking the "Pseudo-Stimulation" option on the screen. After the rising phase, the current will drop directly to 0mA, imitating the sensation of a real stimulation.
  Arms: Sham group

SUMMARY:
This trial is a single-center, single-blind, randomized, sham-stimulation controlled clinical trial. The primary objective of the trial is to detect the targeted effect of tTIS on the nucleus accumbens of adolescent depression patients using functional magnetic resonance imaging (MRI). The secondary objective is to evaluate the potential therapeutic efficacy of TIS treatment for adolescent MDD by assessing changes in clinical characteristics of participants, electrophysiological outcomes, and providing feasibility and tolerance estimates for large-scale efficacy trials. Thirty adolescent MDD participants aged 13 to 17 will be recruited and randomly assigned to receive 10 TIS treatments or sham stimulation treatments (15 participants per group). The trial includes pre-treatment and post-treatment MRI brain scans, clinical assessments, and resting-state EEG, fNIRS acquisition. Follow-ups will be conducted at baseline, after the 10th day of treatment, at the 4th week, and the 8th week. The Montgomery-Åsberg Depression Rating Scale (MADRS), the 17-item Hamilton Depression Rating Scale (HAMD-17), and the Self-Rating Depression Scale (SDS) will be used to assess changes in depressive symptoms of the subjects. The Hamilton Anxiety Rating Scale (HAMA) and the Self-Rating Anxiety Scale (SAS) will be used to assess anxiety symptoms of the subjects. The Wechsler Adult Intelligence Scale-Revised China (WAIS-RC) will be used to assess cognitive function of the subjects.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age 13 - 17 years old; 2)Meet the DSM-5 criteria for MDD with a current MDE without psychotic features, as confirmed by the MINI 3) HAMD-17 total score of ≥20 4) No change in treatment regimen in the 4 weeks prior to screening 5) No severe mental disorders or intellectual disabilities; 6)Can cooperate actively with the experimental process and subsequent follow-up.

Exclusion Criteria:

* 1) serious diseases such as heart, liver, kidney and hematopoietic system disorders; 2) abuse drugs or are addicted to alcohol or suffer from uncontrollable mental illnesses; 3) Active suicidal intent, confirmed by the MINI Module B (Suicidality) or HAMD-17 item #3 score ≥3; 4) Pregnant or lactating; 5) Those who have identified definite organic lesions such as infarction foci, softening foci, hemorrhage foci, and space-occupying lesions through plain scan of cranial MRI; 6) Those with implanted objects in the brain (such as aneurysm clips, shunt devices, stimulators, cochlear implants or electrodes) or any other metal objects in or near the head, and cannot be safely removed; 7) Change in medication or psychotherapy treatment regimen before screening 8) Could not cooperate with fMRI examination or tTIS treatment; 9)Have received other forms of brain stimulation treatment in the past 3 months.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The change in Montgomery-Asberg Depression Rating Scale (MADRS) between groups overtime | baseline, 10 days, 28 days, 56 days
  The change in Montgomery-Asberg Depression Rating Scale (MADRS) between groups overtime